CLINICAL TRIAL: NCT05967247
Title: The Effect of App-Based Mindfulness-Based Stress on Physiological and Psychological Factors in Patients With Heart Failure: A Randomized Controlled Trial
Brief Title: MBSR on Physiological and Psychological Factors in Patients With HF
Acronym: MBSR-PP-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 202307171RINA
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
Keywords: Mindfulness-based stress reduction; Application; Resilience; Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Masking Description: Difficult to blind study caregivers and study outcome assessors due to the nature of the mindfulness-based stress reduction intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR (Experimental): The experimental group used App for MBSR intervention The main app of this experiment is "Mindfulness in life (Taiwan)" (this system is only applicable to Android devices). The content is divided into two parts. The course is compressed and simplified, mainly focusing on mindfulness learning and practising audio-visuals. There are eight-week themed audio-visuals and mindful caring words guided by mindfulness-based stress reduction, mindfulness-stretching guidance, and the function of recording the reading time of the research subjects. App platform for researchers to communicate.
  Interventions: Other: The experimental group used App for MBSR intervention; Other: the "Heart Care Life" app; Other: APP
- waiting list (Placebo Comparator): The waiting list used only the Heart Care Life app for the first eight weeks, as self-management is an essential element of heart failure treatment (Tsami et al., 2023), following the situation-specific theory of heart failure self-management (the situation- specific theory of heart failure self-care:) (Riegel et al., 2022) and American heart failure guidelines (Heidenreich et al., 2022) design (Tsami et al., 2023; Vellone et al., 2020), mainly for Disease-related knowledge and self-management tools, built-in disease health education electronic audiobooks, diet sodium content calculator, diet water content calculator, activity step calculation, etc., to help research subjects self-manage the disease.
  Measure T2 at week 8. From the ninth to the sixteenth week, use the Mindful Live app.
  Interventions: Other: the "Heart Care Life" app; Other: APP

INTERVENTIONS:
Other: The experimental group used App for MBSR intervention — The experimental group used App for MBSR intervention The main app of this experiment is "Mindfulness in Life (Taiwan)" (this system is only applicable to Android devices). The content is divided into two parts. The course is compressed and simplified, mainly focusing on mindfulness learning and practicing audio-visuals. There are eight-week themed audio-visuals and mindful caring words guided by mindfulness-based stress reduction, mindfulness-stretching guidance, and the function of recording the reading time of the research subjects. App platform for researchers to communicate.
  Other Names: Control group serves as a waiting list with priority given to placebo Placebo for the "Heart Care Life" app.
  Arms: MBSR
Other: the "Heart Care Life" app — Control group serves as a waiting list with priority given to placebo Placebo for the "Heart Care Life" app.
Other: APP — APP

SUMMARY:
Objective

The purpose of this study is to explore the relationship between mindfulness, resilience, depression and quality of life in patients with heart failure, and the effect of mindfulness-based stress reduction intervention with mobile phone application on subjects with depressive symptoms. Therefore, the research objectives are as follows:

1. To explore the relationship between mindfulness, resilience, depression, and quality of life in patients with heart failure, and to explore the mediating role of positive emotions (mindfulness, resilience).
2. Using a mobile phone app to conduct mindfulness-based stress reduction interventions, to explore the effects of physiological and psychological factors in heart failure patients with depressive symptoms.

Methods This study will be conducted in two parts. The first part will be a cross-sectional study. It is planned to be conducted in the cardiology ward or outpatient clinic of a university-affiliated hospital in northern Taiwan between September and December 2023 after the approval of the Human Experiment Ethics Committee. Contact the patients who meet the research conditions, adopt the intentional sampling method, and plan to accept 180 research objects for the questionnaire survey, the collection tools are the basic information of the research objects, mindfulness, resilience, depression, quality of life scale; in the first part, the patients' Health Questionnaire (patient health questionnaire-9, PHQ-9) was used to screen for depressive symptoms, and when the total score ≧ 5 points, they were invited to participate in the second part of the study. The second part plans to include 68 subjects in the study, adopting a single-blind random allocation waiting list design, using the app designed by the researcher to implement the mindfulness-based stress reduction intervention program, which is planned to be carried out for 8 weeks, and since the beginning of the study, the 8th week (After the intervention in the experimental group), and the 16th week (after the intervention in the control group), a total of three research data collections were carried out.

DETAILED DESCRIPTION:
Expected research results The expected results of the first part of the research are that the research subjects with higher mindfulness have less depression, higher resilience, and better quality of life, and the mindfulness of the research subjects can play a mediating role between depression and quality of life; the second part expects the research subjects After receiving the intervention of mindfulness-based stress reduction on the mobile phone application, it can increase their mindfulness, resilience and quality of life, reduce depression, blood pressure, and improve heart rate variability.

ELIGIBILITY:
1. Inclusion Criteria:

   * (1) The diagnosis of heart failure is confirmed by a clinician, and the definition of the diagnosis is based on the international statistical classification of diseases and related health problems 10th revision (ICD-10), including I50 Heart failure ( heart failure) related diagnostic codes.
   * (2) Legally recognized as an adult ≧ 18 years old.
   * (3) The second part of the experimental research, in addition to the above inclusion conditions, also needs to have a patient health questionnaire ≥ 5 points, which means mild or above (including) depression (Kroenke et al., 2001; Yeung et al., 2008) can be included in the study.
2. Exclusion Criteria:

   * (1) Diagnosed by a physician as having depression or taking antidepressant drugs regularly, such as selective serotonin reuptake inhibitor (SSRI), serotonin and norepinephrine reuptake inhibitor (serotonin-norepinephrine reuptake inhibitors (SNRI), tricyclic antidepressants (TCA), monoamine oxidase inhibitors (monoamine oxidase inhibitor, MAOI), tetracyclic antidepressants (TeCA), norepinephrine And specific serotonergic antidepressants (Noradrenergic and specific serotonergic antidepressants, NaSSA).
   * (2) New York heart association functional classification (NYHA Fc) IV, which means that it is uncomfortable to perform any physical activity, even when lying in bed or moving, you may feel symptoms such as dyspnea or palpitations.
   * (3) Those who still need to use oxygen or breathing aids throughout the day.
   * (4) Those who are still equipped with ventricular assist devices and rely on life-support devices.
   * (5) Activities of daily living (ADL) < 60 points, unable to take care of themselves in daily life.
   * (6) For those with abnormal cognitive function, the mini-mental state examination (MMSE) < 24 points.
   * (7) Those who have undergone heart transplantation have lost innervation because there is no connection between the autonomic nerve and the heart (McCraty & Shaffer, 2015).
   * (8) In the second part of the interventional experimental research, in addition to the above exclusion conditions, in order to avoid interference with the research, it is also necessary to exclude:
   * A. Those who cannot read traditional Chinese or communicate in Mandarin or Taiwanese, because health education-related materials, videos and applications are all in traditional Chinese.
   * B. Those who cannot use Android devices at home with smartphones or tablets need to operate the application at home due to intervention measures.
   * C. Those who have regularly taken measures related to mindfulness, meditation, and sitting meditation in the past year are not included in order to avoid interfering with the research results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
quality of life (SF-12v2） | T0, T1 = 8 weeks, T2 = 16 weeks.
  short-form health survey (SF-12v2）, Cronbach's α = 0.76～0.85.

SECONDARY OUTCOMES:
depression | T0, T1 = 8 weeks, T2 = 16 weeks.
  patient health questionnaire (PHQ-9）, Cronbach's α = 0.84
mindfulness | T0, T1 = 8 weeks, T2 = 16 weeks.
  five facet mindfulness questionnaire-short form (FFMQ-SF）, Cronbach's α= 0.69～0.85.
Resilience | T0, T1 = 8 weeks, T2 = 16 weeks.
  Connor-Davidson resilience scale (CD-RISC-10）, Cronbach's α = 0.94

OTHER OUTCOMES:
medication adherence | T0, T1 = 8 weeks, T2 = 16 weeks.
  Medication Adherence Self-Reported by Patient
Heart rate variability (HRV) | T0, T1 = 8 weeks, T2 = 16 weeks.
  Measured with a non-plunging wrist-worn instrument
heart rate (pulse) | T0, T1 = 8 weeks, T2 = 16 weeks.
  Measured according to the blood pressure measuring instrument regularly calibrated by the hospital
blood pressure (BP) | T0, T1 = 8 weeks, T2 = 16 weeks.
  Measured according to the blood pressure measuring instrument regularly calibrated by the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] MIT (2012). APP Inventor. Massachusetts Institute of Technology. United States. https://appinventor.mit.edu/
- [Background] Edhouse J, Wardrope J, Morris FP. Call to needle times after acute myocardial infarction. Delay in calling for help for chest pain. BMJ. 1999 Feb 27;318(7183):597; author reply 598. No abstract available. PMID 10037647
- [Background] Riegel B, Dickson VV, Vellone E. The Situation-Specific Theory of Heart Failure Self-care: An Update on the Problem, Person, and Environmental Factors Influencing Heart Failure Self-care. J Cardiovasc Nurs. 2022 Nov-Dec 01;37(6):515-529. doi: 10.1097/JCN.0000000000000919. Epub 2022 Apr 27. PMID 35482335
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):e263-e421. doi: 10.1016/j.jacc.2021.12.012. Epub 2022 Apr 1. PMID 35379503
- [Background] McCraty R, Shaffer F. Heart Rate Variability: New Perspectives on Physiological Mechanisms, Assessment of Self-regulatory Capacity, and Health risk. Glob Adv Health Med. 2015 Jan;4(1):46-61. doi: 10.7453/gahmj.2014.073. PMID 25694852
- [Background] Vandenbogaart E, Gawlinski A, Grimley KA, Lewis MA, Pavlish C. App-Based Mindfulness Intervention to Improve Psychological Outcomes in Pretransplant Patients With Heart Failure. Crit Care Nurse. 2023 Apr 1;43(2):15-25. doi: 10.4037/ccn2023411. PMID 37001879
- [Background] Tabernero C, Gutierrez-Domingo T, Steca P, Castillo-Mayen R, Cuadrado E, Rubio SJ, Farhane-Medina NZ, Luque B. Effectiveness of Mindfulness and Positive Strengthening mHealth Interventions for the Promotion of Subjective Emotional Wellbeing and Management of Self-Efficacy for Chronic Cardiac Diseases. J Pers Med. 2022 Nov 25;12(12):1953. doi: 10.3390/jpm12121953. PMID 36556174
- [Background] MacEwen EG, Brown NO, Patnaik AK, Hayes AA, Passe S. Cyclic combination chemotherapy of canine lymphosarcoma. J Am Vet Med Assoc. 1981 Jun 1;178(11):1178-81. No abstract available. PMID 6895078
- [Background] Heo S, McSweeney J, Ounpraseuth S, Shaw-Devine A, Fier A, Moser DK. Testing a Holistic Meditation Intervention to Address Psychosocial Distress in Patients With Heart Failure: A Pilot Study. J Cardiovasc Nurs. 2018 Mar/Apr;33(2):126-134. doi: 10.1097/JCN.0000000000000435. PMID 28661991
- [Background] Curtis PJ. Globin mRNA in Friend cells: its structure, function and synthesis. Biochim Biophys Acta. 1980 Sep 22;605(3):347-64. doi: 10.1016/0304-419x(80)90016-5. PMID 6996728
- [Background] Simas W, Chiossi JC, Abib OA. [Urethral prolapse in a young woman]. Rev Paul Med. 1972 Aug;80(2):83-6. No abstract available. Portuguese. PMID 4671576
- [Background] Kang Q, Luo A. The efficacy of mindfulness-based intervention for heart diseases: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2022 Sep 30;101(39):e29649. doi: 10.1097/MD.0000000000029649. PMID 36181030
- [Background] Jalali D, Abdolazimi M, Alaei Z, Solati K. Effectiveness of mindfulness-based stress reduction program on quality of life in cardiovascular disease patients. Int J Cardiol Heart Vasc. 2019 Apr 12;23:100356. doi: 10.1016/j.ijcha.2019.100356. eCollection 2019 Jun. PMID 31011624
- [Background] Baumel A, Muench F, Edan S, Kane JM. Objective User Engagement With Mental Health Apps: Systematic Search and Panel-Based Usage Analysis. J Med Internet Res. 2019 Sep 25;21(9):e14567. doi: 10.2196/14567. PMID 31573916
- [Background] Felsted KF. Mindfulness, Stress, and Aging. Clin Geriatr Med. 2020 Nov;36(4):685-696. doi: 10.1016/j.cger.2020.06.010. Epub 2020 Aug 17. PMID 33010903
- [Background] Kabat-Zinn, J., & Hanh, T. N. (2009). Full catastrophe living: Using the wisdom of your body and mind to face stress, pain, and illness. Delta.
- See also: Chih-fan Yeh — https://orcid.org/0000-0002-0678-2264
- See also: Chia-Jung Hsieh — https://orcid.org/0000-0002-1062-8307
- See also: Shu-Ling Wang — https://orcid.org/0000-0002-4336-765X